CLINICAL TRIAL: NCT03597009
Title: A Phase Ib/II Study of IV Nivolumab and Intrapleural Talimogene Laherparepvec for Patients With Malignant Pleural Effusion
Brief Title: A Study of Nivolumab and Intrapleural Talimogene Laherparepvec for Malignant Pleural Effusion
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to slow accrual and withdrawal of funding
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: C. R. Bard (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1626
Record Dates: First submitted 2018-06-01; First posted 2018-07-24 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Malignant Pleural Effusion; Stage IV Metastatic Cancer; Lung Cancer
Keywords: talimogene laherparepvec; Nivolumab; PleurX
MeSH Terms: conditions — Pleural Effusion, Malignant; Neoplasm Metastasis; Lung Neoplasms | interventions — talimogene laherparepvec; Nivolumab

STUDY DESIGN:
Intervention Model Description: We will conduct a Phase Ib/II trial that includes a safety run-in period using 3 +3 dose escalation rules to evaluate the feasibility of administering talimogene laherparepvec into the intrapleural space of subjects with malignant pleural effusion (MPE) via a pleurX catheter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label, single-arm Phase I (Experimental): Talimogene laherparepvec (TVEC) administered into the intrapleural space of subjects with malignant pleural effusion (MPE) via a pleurX catheter with or without nivolumab
  Interventions: Drug: Talimogene laherparepvec (TVEC); Drug: Nivolumab

INTERVENTIONS:
Drug: Talimogene laherparepvec (TVEC) — Talimogene laherparepvec (TVEC) (4ml of 108 pfu/ml) for up to 9 cycles, with or without nivolumab
  Other Names: Imlygic; OncoVex
Drug: Nivolumab — Nivolumab (240 mg IV) will be co-administered with talimogene laherparepvec (TVEC) (4ml of 108 pfu/ml) for up to 9 cycles in the Dose Level 2 cohort
  Other Names: Opdivo

SUMMARY:
This is a Phase Ib/II clinical trial to evaluate the feasibility of administering talimogene laherparepvec into the intrapleural space of subjects with malignant pleural effusion through a pleurX catheter.

DETAILED DESCRIPTION:
This is a phase 1b/II clinical trial that includes a safety run-in cohort to investigate the novel approach of administering intrapleural talimogene laherparepvec via a pleurX catheter in patients with known malignant pleural effusion (MPE).

In Phase Ib of this study, the safety of infusing talimogene laherparepvec directly into the pleural cavity of subjects diagnosed with MPE, through pleurX catheter, will be tested.

In Phase II of this study, after establishing the safety of the above mentioned approach, 24 subjects will enrolled and treated with intrapleural talimogene laherparepvec and IV nivolumab.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria to participate in this study:

1. Be ≥ 18 years of age on day of signing informed consent.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
3. Histologically or cytologically confirmed stage IV metastatic cancer.
4. Confirmation of malignant pleural effusion via imaging (Computer tomography (CT) scan, chest x-ray (CXR), MRI, ultrasound, Positron Emission Tomography (PET)/CT), and cytology for which pleurX catheter placement is standard of care
5. Recovered from all reversible toxicities related to their previous treatment (other than alopecia) to ≤grade 1 or baseline; exceptions to this criterion may be allowed following review by the principal investigator for toxicities that are not expected to be exacerbated by nivolumab or talimogene laherparepvec. Grade 2 peripheral neuropathy will not result in exclusion as neither study agent would be expected to exacerbate it.
6. No history of untreated brain metastasis. Treated brain metastases must not be known to be progressive, symptomatic, or currently requiring > 10 mg of prednisone or prednisone equivalents within two weeks prior to study drug administration.
7. Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication. Females of childbearing potential must agree to use 2 methods of effective contraception or abstain from heterosexual sex throughout the treatment period and for 5 months after the last dose of study treatment. Females of childbearing potential are women who have not been surgically sterilized (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or have not been free of menses for >1 year.
8. Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e. double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 7 months after the last dose of study treatment.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria will not be able to participate in this study:

1. Receiving any investigational agent, or using an investigational device, currently or within 28 days or 5 half-lives of Day 1 of treatment on this study, whichever is longer.
2. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1, or who has not recovered to, ≤ Grade 1 toxicity at baselines from adverse events due to agents administered more than 4 weeks earlier. Exceptions to these criteria may be allowed at the discretion of the investigator for toxicities that are not expected to be exacerbated by nivolumab or talimogene laherparepvec (e.g., alopecia, peripheral neuropathy, etc).
4. Has received prior therapy with an anti-programmed cell death receptor (PD)-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
5. Any concurrent chemotherapy, intraperitoneal (IP), biologic or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
6. Major surgery within 28 days prior to day 1 of study treatment from which the patient has not completely recovered.
7. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
8. Has a known secondary malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
9. Has a history of non-infectious pneumonitis that required steroids; currently active non-infectious pneumonitis; or evidence of interstitial lung disease.
10. Has an active infection requiring systemic therapy or history of uncontrolled infection.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. This includes known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial. This also includes unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction ≤ 6 months prior to study entry.
12. Has inadequate home environment or social support to safely complete the trial procedures
13. Is pregnant or breastfeeding
14. Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or evidence of active hepatitis B virus (HBV).
15. Has a multi-loculated pleural effusion that would not lead to relief of dyspnea from drainage of a single loculation.
16. Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
17. Active herpetic skin lesions or prior complications of herpetic infection or requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
18. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina (UNC) Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials//clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between March 2019 and August 2020.
Period: Overall Study
Arm/Group | Open-label, Single-arm Phase I
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I Number of Participants With Treatment-related Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by the NCI Common Terminology Criteria for Adverse Events which is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: from day 1 of treatment to 30 days after the last dose of study medication (approximately 11 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Phase II Resolution of MPE
Description: The rate of resolution of malignant pleural effusion following IV nivolumab combined with intrapleural injection of talimogene laherparepvec
Time Frame: 13 weeks
Population: No participants were enrolled on the Phase II portion of the study
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival from day 1 of treatment until death or progression. Per immune-related Response Evaluation Criteria in Solid Tumours (irRECIST), immune-related Progressive Disease (irPD)is defined as at least 20% and minimum 5 mm absolute increase in total measured tumor burden compared to nadir, or irPD for non-target or new un-measurable lesions.
Time Frame: up to 2 years
Measure: Number; unit: days
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 1
days | 85

4. Secondary Outcome: Overall Survival
Description: Overall survival from day 1 of treatment until death
Time Frame: up to 2 years
Measure: Number; unit: days
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 1
days | 85

5. Secondary Outcome: Response Rate
Description: Response rate after treatment per Immune-Related Response Evaluation Criteria In Solid Tumors (irRECIST) defined as the proportion of patients with reduction in tumor (immune-related Complete Response (irCR) or immune-related Partial Response (irPR)). irCR is a complete disappearance of all lesions (whether measurable or not) and no new lesions. Lymph nodes must decrease to <10mm in short axis. irPR is a decrease in tumor burden ≥ 30%, in total measured tumor burden relative to baseline, non-target lesions are not in complete response (disappearance of all lesions) and not unequivocal progression or new non-measurable lesions.
Time Frame: up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 1
proportion of participants | 0

6. Secondary Outcome: Phase II Number of Participants With Treatment-related Adverse Events
Description: as for outcome 1
Time Frame: 13 weeks
Population: No participants were enrolled in the Phase II portion of the study
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 0

7. Secondary Outcome: Average Dyspnea Score
Description: Results from patient reports of the Modified Borg Scale of Perceived Dyspnea, measuring change in scale over time. The scale evaluates perceived level of shortness of breath ranging from 0 to 10, where 0 indicates the greatest success of the treatment.
Time Frame: 13 weeks
Measure: Number; unit: score on a scale
Arm/Group | Open-label, Single-arm Phase I
Number analyzed (Participants) | 1
score on a scale | 4

ADVERSE EVENTS:
Time Frame: From day one of treatment to 30 days after the last dose of treatment (approximately 11 weeks)
Arm/Group | Open-label, Single-arm Phase I
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Single-arm Phase I (N=1)
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Single-arm Phase I (N=1)
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Fever (General disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Study terminated early due to slow accrual and withdrawal of funding so only one participant was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03597009/Prot_SAP_000.pdf